CLINICAL TRIAL: NCT01348425
Title: Evaluation of the Zilver PTX Drug-Eluting Peripheral Stent
Brief Title: Zilver PTX Drug-Eluting Peripheral Stent Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-003
Record Dates: First submitted 2011-04-29; First posted 2011-05-05 (Estimated); Results first posted 2014-04-16 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2014-03

CONDITIONS: Peripheral Arterial Disease
Keywords: PAD
MeSH Terms: conditions — Peripheral Arterial Disease

ARMS (2):
- Longer Stents (Experimental)
  Interventions: Device: Longer Zilver PTX Stents
- Shorter Stents (Experimental)
  Interventions: Device: Shorter Zilver PTX Stents

INTERVENTIONS:
Device: Longer Zilver PTX Stents — Treatment with at least one 100 mm or longer Zilver PTX stent
  Arms: Longer Stents
Device: Shorter Zilver PTX Stents — Treatment with Zilver PTX stents 80 mm or shorter only
  Arms: Shorter Stents

SUMMARY:
This randomized, post-market clinical study is intended to evaluate the delivery and deployment of longer Zilver PTX stents (≥ 100 mm) compared to shorter Zilver PTX stents (≤80 mm) for treatment of lesions of the above-the-knee femoropopliteal artery.

ELIGIBILITY:
Inclusion Criteria:

* One de novo or restenosed artherosclerotic lesion with > 50% diameter stenosis
* Reference vessel diameter of 4 - 9 mm
* Rutherford category ≥ 2
* Resting ankle brachial index < 0.9

Exclusion Criteria:

* Prior stent in the study vessel
* Significant stenosis (> 50%) or occlusion of inflow tract not successfully treated before the study procedure
* Lacks at least one patent runoff vessel
* Lesions requiring atherectomy, cutting balloons, cryoplasty balloons, or any other advanced device to facilitate stent delivery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-05; Primary Completion 2011-10 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. med. Jens Ricke, Principal Investigator — Universitätsklinikum Magdeburg A.ö.R., Department for Radiology and Nuclear Medicine
Locations (4):
- Germany (3):
  - Herz-Zentrum, Bad Krozingen
  - Evangelische Krankenhaus Königin Elisabeth Herzberge, Berlin
  - Universitätsklinikum Magdeburg A.ö.R., Magdeburg
- INSELSPITAL, Universitätsspital Bern, Bern, Switzerland

RESULTS

PARTICIPANT FLOW:
Groups:
- Longer Stents: Longer Zilver PTX Stents : Treatment with at least one 100 mm or longer Zilver PTX stent
- Shorter Stents: Shorter Zilver PTX Stents : Treatment with Zilver PTX stents 80 mm or shorter only
Period: Overall Study
Arm/Group | Longer Stents | Shorter Stents
Started | 31 | 14
Completed | 30 | 13
Not Completed | 1 | 1
Not completed — Imaging was not taken. | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Longer Stents | Shorter Stents | Total
Number analyzed (Participants) | 31 | 14 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (9.2) | 71.6 (8.3) | 68.8 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 23 | 9 | 32

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Stent Length Upon Deployment
Time Frame: During Procedure (day 1) (Prior to Stent Deployment and after Stent Deployment)
Measure: Mean (Standard Deviation); unit: Change in stent length (%)
Arm/Group | Longer Stents | Shorter Stents
Number analyzed (Participants) | 30 | 13
Change in stent length (%) | 0.5 (4.2) | -0.2 (3.8)
Statistical Analysis 1: Comparison: Longer Stents vs Shorter Stents; The alternative hypothesis is equivalence in mean change in stent length upon deployment between longer and shorter stents, i.e., the difference in mean change between the longer and shorter stents is close to 0. Thus, a small p-value indicates a 95% confidence interval covers 0; Test type: Non-Inferiority or Equivalence — The equivalence margin is +/- 10%, type I error is assumed to be 0.05, with a power of 0.8; p < 0.01, t-test, 2 sided — Schuirman's TOST equivalence test on change in stent length upon deployment between longer and shorter stents; To test the hypothesis whether the percent change in stent length is contained within [-10%, 10%]; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-2.0 to 3.5], Standard Deviation 4.1

ADVERSE EVENTS:
Time Frame: 30 days
Groups:
- Stented Patients: The adverse events were combined because all patients were treated with Zilver PTX stents. The safety of Zilver PTX has been previously established and the primary objective of this study was changes in post-deployment stent length; i.e. immediately post-procedure.
Arm/Group | Stented Patients
Serious Adverse Events (participants affected / at risk) | 5/45
Other Adverse Events (participants affected / at risk) | 0/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stented Patients (N=45)
Renal disease (Renal and urinary disorders) | 1 (1) — failed hemodialysis shunt requiring revision (Due to a pre-existing condition.)
Pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) — exacerbation of COPD (Due to a pre-existing condition.)
Orthopedic/vascular repair (Surgical and medical procedures) | 1 (1) — lumbar protrusion (Due to other medical problems.)
Restenosis/occlusion of study lesion (Vascular disorders) | 1 (1)
Restenosis/occlusion of non-study limb (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days